CLINICAL TRIAL: NCT07081880
Title: Study of the Pathophysiological Mechanisms Involved in the SAPHO Syndrome: Genetic Component and Immune Response
Acronym: SAPHO-Screen
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 644_SAPHO-Screen
Record Dates: First submitted 2025-06-18; First posted 2025-07-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: SAPHO Syndrome
MeSH Terms: conditions — Acquired Hyperostosis Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- biological sampling
  Interventions: Other: biological sampling

INTERVENTIONS:
Other: biological sampling — DNA and Cells will be sampled

SUMMARY:
SAPHO syndrome (Synovitis, Acne, Pustulosis, Hyperostosis and Osteitis) is a chronic inflammatory rheumatism associating bone or joint lesions and dermatological manifestations dominated by severe acne and palmar and palmoplantar pustulosis. Prevalence of SAPHO syndrome is estimated at 1/50000 in France, but this figure is probably underestimated due to frequent misdiagnosis. Osteoarticular manifestations form a rheumatic picture very similar to that of other forms of spondyloarthritis (SpA). The latest French recommendations do not distinguish SAPHO syndrome from other forms of SpA. As a result, the management of SAPHO remains fairly heterogeneous, essentially based on the local experience of rheumatologists. Delays in diagnosis and difficulties in finding effective treatment can result in significant disability and reduced quality of life, particularly detrimental in a young population (age at diagnosis is usually between 30 and 40). The wide spectrum of clinical presentations of SAPHO syndrome explains the complexity of managing this condition. Understanding the pathophysiological mechanisms underlying these different forms of the disease is a major challenge for personalized medicine. SAPHO syndrome is a multifactorial disease that is a result of interaction of genetic, environmental, immunological and infectious factors. In the classification of immune-mediated inflammatory diseases, SAPHO syndrome lies midway between autoinflammatory diseases involving the innate immune response and spondyloarthritis associated with abnormalities in the adaptive immune response. Indeed, while the clinical phenotype may resemble spondyloarthritis in certain aspects, the identification of genetic forms of chronic relapsing osteitis, such as DIRA syndrome or Majeed syndrome, argues in favor of an autoinflammatory origin of SAPHO syndrome. Although osteitis is reputed to be sterile, an infectious initiating factor has long been suspected in this disease. Among the bacterial agents, antigens antigens from Cutibacterium acnes were detected in bone biopsies from patients with SAPHO syndrome. It has been suggested that this bacterium may play a role in triggering a systemic inflammatory response systemic inflammatory response mediated in particular by IL-1β.

DETAILED DESCRIPTION:
Although neutrophils (PNN) are the most abundant leukocytes in the circulation and form a first line of innate immune defense, they are difficult to study because they have a short lifespan and, after migrating into tissues, are rapidly eliminated by macrophages. PNN play a central role in the early phase of SpA development, and contribute to the various tissue damage observed. PNN are recruited from the circulation and enter target tissues such as joints, enthesis, digestive tract, skin and eyes, where they produce neutrophil extracellular traps (NETs), cytokines and chemokines that attract other immune cells. In SAPHO syndrome, bone biopsy usually reveals an infiltrate of PNNs, at least in the early stages of the disease. To date, no study has performed extensive phenotyping of circulating blood to identify over- or under-represented cell populations, which could thus be implicated in the disease.

Studies showed an increase in the Th17 population in SAPHO patients, elevated low density granulocytes and neutrophil extracellular traps formation, as well as specific protein patterns associated with inflammation. Genetic studies, particularly in Chinese populations, have revealed potential associations with IL-23R and IL-4 genes, as well as SNPs in PEX16 and IQCA1L. However, no large-scale genetic analysis has been conducted in European/Caucasian populations. While certain forms of SAPHO syndrome suggest a genetic predisposition, studies targeting genes associated with monogenic disorders like Majeed, PAPA, and DIRA have yielded negative results. Chinese studies have indicated involvement of genes like CSF2RA, NOD2, MEGF6, and ADAM5. Despite genetic predisposition suspicions, robust associations have not been identified, particularly in Caucasian populations, warranting further research.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient diagnosed with SAPHO syndrome
* Weight > 35 kg
* Patient affiliated with a health insurance plan
* French-speaking patient
* Patient who has given free, informed, and written consent

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient diagnosed with SAPHO syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2035-05-15 (Estimated)

PRIMARY OUTCOMES:
Investigating a Genetic Predisposition to SAPHO Syndrome | at baseline
  Comparison of allelic frequencies in patients with SAPHO syndrome versus the general population

SECONDARY OUTCOMES:
Estimating the Degree of Genetic Component Overlap Between SAPHO Syndrome and Axial SpA | at baseline
  Comparison of allelic frequencies in patients with SAPHO syndrome versus patients with severe and non-severe axial SpA
Studying the Genetic Component Based on Different Phenotypes of SAPHO Syndrome | at baseline
  comparison of allelic frequencies among patients:
  With pure osteitis form of SAPHO syndrome vs. those with axial form of the disease With cutaneous involvement vs. without cutaneous involvement
Studying the Functional Consequences of Variants Associated with SAPHO Syndrom, on the protein level | at baseline, at 6 months, and every year for 9 years
  comparison of Expression level of protein of the different variants in sorted cells and plasma
Studying the Functional Consequences of Variants Associated with SAPHO Syndrom, on the transciptom level | at baseline, at 6 months, and every year for 9 years
  comparison of Expression level of mRNA of the different variants in sorted cells and plasma
Phenotypic Characterization of Different Circulating Immune Subpopulations in Patients with SAPHO Syndrome | at baseline and at 6months
  percentage of the different circulating immune cell subtypes (monocytes, T lymphocytes and subclasses, B lymphocytes, PNN, and NK) and rare populations (MAIT, γδ lymphocytes, etc.) determined by flow cytometry techniques
Measurement of Cytokines of Interest | at baseline and at 6months
  Dosage of cytokine done by ELISA in the plasma of SAPHO patients and control populations.
Identification of Prognostic Factors for Severity of SAPHO Syndrome and/or Response to Different Treatments | at baseline and at 6months
  clinical evalution of the severity of the disease and its response to the treatment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Cochin, Paris
  - Hôpital Paris Saint Joseph, Paris

IPD SHARING:
Plan to Share IPD: No